CLINICAL TRIAL: NCT07068061
Title: Evaluation of the Performance and Safety of Polydioxanone Suture (PDO) "Bio Meyisun" for the Temporary Correction of the Mid-face Area.
Brief Title: PER-SAF_PDOS (Performance and Safety of Polydioxanone Suture)
Acronym: PER-SAF_PDOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 21 Century Medical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-MD-CIP-004
Record Dates: First submitted 2025-06-27; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Wrinkles; Anti Aging; Face-lift

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional arm (Experimental): The procedure will start with skin cleansing using an antiseptic and careful marking of entry and exit points for thread placement. Aesthetic cream and local anaesthesia will be applied to enhance patient comfort before inserting PDO barbed threads into the subdermal layer using a cannula. The threads will be adjusted to create a natural-looking lift, followed by manual lifting to anchor them securely within the tissue. Finally, any excess thread will be trimmed, the area massaged for proper positioning, and the skin cleaned again to maintain sterility.
  Interventions: Device: PDO suture

INTERVENTIONS:
Device: PDO suture — A biodegradable polymer used in dissolvable sutures and lifting threads, stimulating collagen production as it degrades.

SUMMARY:
This clinical investigation aims to confirm the safety and efficacy of the ID in facial soft tissue reconstruction, specifically for non-incision surgery to tighten and lift the facial skin for a rejuvenated facial appearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old with full legal capacity, male and female;
* Patients with ability to understand the proposed aesthetic correction and to understand and sign informed consent;
* Patients who are willing and able to comply with scheduled visits, aesthetic correction procedure and other trial procedures.

Exclusion Criteria:

* Pregnant or breast--feeding women;
* Patients currently participating in any other clinical investigation;
* Patients who have received a vaccine within 14 days prior to the baseline or plan to have vaccine within 14 days after the injection;
* Patients with a medical history of systemic diseases, including severe kidney, liver, heart and neurological disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
The assessment of improvement in mid-face appearance. | up to 24 weeks
  Proportion of subjects with any improvement compared to baseline, as assessed by the Independend Evaluator (IE).

SECONDARY OUTCOMES:
Further evaluation of improvement of the mid-face appearance. | up to 35 weeks
  Proportion of subjects with any improvement compared to baseline, as assessed by the Independend Evaluator (IE).
Self-evaluation of improvement of the mid-face appearance by the Subject. | up to 35 weeks
  Proportion of subjects with any improvement compared to baseline, as assessed by the Subject.
Number of (S)AEs. | up to 35 weeks
  Number of (S)AEs evaluated by the subject using patient diary